CLINICAL TRIAL: NCT04354688
Title: A Prospective, Randomized, Comparative Clinical Study of the Safety, Efficacy and Clinical Benefits of the T3 Certain Tapered With DCD Implant System
Brief Title: T3 Certain Tapered With DCD vs T3 Certain Tapered Non-DCD
Acronym: Apple
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1802
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: Test implant- T3 Certain Tapered implant with DCD Active Comparator- T3 Certain Tapered implant without DCD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- T3 Certain Tapered implant with DCD (Experimental): Implant will be placed in the maxilla or mandible in a single stage manner and loaded with prosthesis after 6 weeks of healing. Final restorations will take place no later than 4 months following implant placement surgery. The implants will be evaluated yearly for 2 years.
  Interventions: Device: T3 Certain Tapered Implant
- T3 Certain Tapered implant without DCD (Active Comparator): Implant will be placed in the maxilla or mandible in a single stage manner and loaded with prosthesis after 6 weeks of healing. Final restorations will take place no later than 4 months following implant placement surgery. The implants will be evaluated yearly for 2 years.
  Interventions: Device: T3 Certain Tapered Implant

INTERVENTIONS:
Device: T3 Certain Tapered Implant — Patients will be randomized to receive either the T3 Certain Tapered with DCD (Test) or the T3 Certain Tapered without DCD (control/active comparator). Both types of implants will be rehabilitated in the same manner (early loading)

SUMMARY:
This will be a prospective, randomized multicenter study to determine the safety and efficacy of the T3 Certain Tapered with DCD as compared to T3 Certain Tapered without DCD. All implants will be placed in the maxilla or mandible in a single stage manner and loaded with prosthesis after 6 weeks of healing. Final restorations will take place no later than 4 months following implant placement surgery. The implants will be evaluated yearly for 2 years.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized study that will assess the the safety and efficacy of the implant systems with:

* Resistance to countertorque testing (mobility)
* Implant Stability Quotient (ISQ)
* Changes in peri-implant crestal bone levels
* Confirmation of clinical benefits

A total of 60 implants, 30 per treatment group will be placed across all participating sites. One patient may contribute more than 1 implant. All implants/ patients will be followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex and greater than 18 years of age
2. Patients for whom a decision has already been made to use a dental implant in the mandible or maxilla.
3. Immediate extraction or a prior extracted site
4. Patients must be physically able to tolerate conventional surgical and restorative procedures.
5. Presence of opposing dentition
6. Patients who provide a signed informed consent.
7. Patients who agree to be evaluated for each study visit.
8. Minimum primary stability, insertion torque > 35Ncm

Exclusion Criteria:

1. Patients with known systemic diseases such as uncontrolled diabetes, endocrine disease, heart disease, immuno-compromised, or mental disorders.
2. Patients with current use of non-steroidal anti-inflammatory drugs, bisphosphonates or corticosteroid treatments.
3. Patients with active infection or severe inflammation in the areas intended for implant placement.
4. Patients with a > 10 cigarette per day smoking habit.
5. Patients with a history of therapeutic radiation to the head or jaw.
6. Patients who are known to be pregnant at the screening visit or planning to become pregnant within 6 months of study enrollment.
7. Patients with evidence of severe parafunctional habits such as bruxing or clenching.
8. Patients with HIV or Hepatitis infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Implant survival | 2 years
  Assessed by lack of mobility, resistance to countertorque testing, implant stability measurement

SECONDARY OUTCOMES:
Peri-implant crestal bone levels | 2 years
  Assessed by radiographic measurements of serial crestal bone levels

CONTACTS AND LOCATIONS:
Locations (2):
- Hospital San Jose, Providencia, Santiago Metropolitan, Chile
- Dr. George Papavasiliou, Athens, Greece

IPD SHARING:
Plan to Share IPD: No